CLINICAL TRIAL: NCT01368510
Title: Cognitive-Behavioral Therapy and Glutamate in Cingulate Gyrus in OCD
Brief Title: Intensive Cognitive-Behavioral Therapy For Obsessive-Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joseph O'Neill, PhD, Prof Child Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH085900 (NIH); R01MH085900 (NIH)
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
Keywords: obsessive-compulsive disorder (OCD); cognitive-behavioral therapy (CBT); magnetic resonance spectroscopy (MRS); glutamate; cingulate gyrus
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- OCD Active CBT (Experimental): Adults with obsessive-compulsive disorder (OCD) will be treated with cognitive-behavioral therapy (CBT) from the time of enrollment.
  Interventions: Behavioral: Intensive Cognitive Behavioral Therapy (CBT)
- OCD Waitlist (Active Comparator): Adults with OCD will receive waitlist treatment at enrollment. Nonresponders will cross over to CBT.
  Interventions: Behavioral: Intensive Cognitive Behavioral Therapy (CBT); Behavioral: Waitlist
- Healthy Control (No Intervention): Healthy control adults will be given no intervention.

INTERVENTIONS:
Behavioral: Intensive Cognitive Behavioral Therapy (CBT) — Nondrug psychotherapy administered daily 5 days/week for 4 weeks
  Other Names: Exposure and Response Prevention (ERP)
  Arms: OCD Active CBT; OCD Waitlist
Behavioral: Waitlist — Minimal contact waitlist weekly for 4 weeks
  Arms: OCD Waitlist

SUMMARY:
Even with the best available treatments for obsessive-compulsive disorder (OCD), most patients only partially recover and many patients do not respond at all. Such incomplete and inadequate response contributes to greater public health costs in terms of morbidity and patient care expenses. This study aims for a better understanding of abnormal brain chemistry in OCD and how it is affected by cognitive-behavioral therapy (CBT) in order to develop novel therapies and improve the success of existing therapies. The main hypothesis is that CBT will change levels of the excitatory neurotransmitter glutamate in OCD patients in a region of the brain involved in OCD known as the cingulate cortex.

DETAILED DESCRIPTION:
This study will characterize the neurochemical abnormalities in important brain circuits underlying obsessive-compulsive disorder (OCD) symptoms and the effects of cognitive-behavioral therapy (CBT). Identification of such metabolite biomarkers will provide an important foundation for translational clinical studies to maximize the ability of CBT to reduce symptoms and to design medications that target core features of the disease, which is particularly important for those who do not respond to, or have access to, CBT.

OCD is an often disabling and chronic psychiatric condition that affects approximately 2% of the world's population. Most patients respond only incompletely to current treatments and many do not respond at all. CBT, a form of psychotherapy, is one of the most effective treatments for OCD, yet its mechanism of action is not fully understood. The objective of this study is to use neuroimaging to understand how neurometabolite abnormalities in neural circuits relate to OCD symptoms, and how these are affected by CBT. In OCD, dysfunction is suspected in several subregions of the cingulate gyrus, a brain region involved in relevant neural circuits. This study will use magnetic resonance spectroscopic imaging (MRSI) to measure concentrations of brain metabolites, including glutamate (Glu), in the cingulate. Glu is an important excitatory neurotransmitter that is suspected to be disturbed in OCD. In this study, MRSI scans will be performed on 25 adult OCD patients before and after 4 weeks of daily CBT. They will be compared to 25 untreated healthy controls scanned 4 weeks apart. A third group of 25 OCD patients will be scanned before and after 4 weeks while on the waitlist, will then receive 4 weeks of CBT, and will be scanned a third time at its completion. The specific aims of this study are: 1) Determine if levels of the Glu in the "emotional" and "cognitive" subregions of the cingulate differ between OCD patients and controls; 2) Determine if Glu changes after CBT or waitlist in the OCD patients and if they change in the controls after simple passage of time; 3) Determine if there are relationships between Glu and clinical and neurocognitive symptoms of OCD before and after CBT.

ELIGIBILITY:
Inclusion Criteria:

* meets DSM-IV-TR diagnostic criteria for OCD as primary (most severe) diagnosis based on Anxiety Disorders Interview Schedule (ADIS) Clinical Severity Rating
* reported DSM-IV-TR-threshold OCD symptom onset age 18 or later
* Yale-Brown Obsessive-Compulsive total score greater than or equal to 16
* fluent English speaker
* signed informed consent

Exclusion Criteria:

* IQ of less than 80 on the Wechsler Abbreviated Scales of Intelligence
* lifetime DSM-IV diagnosis of pervasive developmental disorder, mania, psychosis, conduct disorder, or substance dependence assessed through ADIS
* current DSM-IV diagnosis of major depressive disorder if ADIS CSR rating is 4 or higher (severe) or attention-deficit hyperactivity disorder
* primary compulsive hoarding
* any changes (dose or agent) in psychotropic medication for OCD or other psychiatric condition within 12 weeks prior to enrollment
* severe illness that requires immediate inpatient psychiatric intervention
* any serious psychiatric, psychosocial, or neurological condition requiring immediate treatment other than that provided in the current study
* any body metal (other than dental fillings), positive pregnancy test, or other MR scan contraindications
* prior trial of CBT for OCD, regardless of outcome
* medical conditions that affect cerebral metabolism (e.g., thyroid disorders or diabetes)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
MRSI glutamate | 4 weeks
  Regional concentration of glutamate in brain, as measured by magnetic resonance spectroscopic imaging (MRSI)

SECONDARY OUTCOMES:
Y-BOCS | 4 weeks
  Severity of core obsessive-compulsive clinical symptoms as measured with the Yale-Brown Obsessive-Compulsive Scale score

CONTACTS AND LOCATIONS:
Overall Officials: Joseph O'Neill, PhD, Principal Investigator — UCLA Child Psychiatry
Locations (1):
- UCLA Obsessive-Compulsive Disorder Intensive Treatment Program, Los Angeles, California, United States

REFERENCES:
- [Derived] Reggente N, Moody TD, Morfini F, Sheen C, Rissman J, O'Neill J, Feusner JD. Multivariate resting-state functional connectivity predicts response to cognitive behavioral therapy in obsessive-compulsive disorder. Proc Natl Acad Sci U S A. 2018 Feb 27;115(9):2222-2227. doi: 10.1073/pnas.1716686115. Epub 2018 Feb 12. PMID 29440404
- [Derived] Moody TD, Morfini F, Cheng G, Sheen C, Tadayonnejad R, Reggente N, O'Neill J, Feusner JD. Mechanisms of cognitive-behavioral therapy for obsessive-compulsive disorder involve robust and extensive increases in brain network connectivity. Transl Psychiatry. 2017 Sep 5;7(9):e1230. doi: 10.1038/tp.2017.192. PMID 28872637